CLINICAL TRIAL: NCT06739941
Title: A Direct-to-Consumer, Open-label Study Investigating the Tolerability of BG-OS in Healthy Individuals in a Home Setting
Brief Title: Investigating the Tolerability of Oat Fiber (BG-OS) in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: One Bio Inc. (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00074413
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Digestive Health; Metabolic Health
Keywords: oat fiber; dietary fiber; beta-glucan; Gastrointestinal tolerability; oat oligosaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5 g/day of oat fiber (Active Comparator): Participants receive 5 g/day of oat fiber (BG-OS) in a single dose
- 10 g/day of oat fiber (Active Comparator): Participants receive 10 g/day of oat fiber (BG-OS) in a single dose.
  Interventions: Other: Oat fiber (BG-OS)
- 20 g/day of oat fiber (Active Comparator): Participants receive 20 g/day of oat fiber (BG-OS) in a single dose.
  Interventions: Other: Oat fiber (BG-OS)

INTERVENTIONS:
Other: Oat fiber (BG-OS) — Beta-glucan oligosaccharide (BG-OS) is beta-glucan predominant, dietary fiber obtained by extracting oat fiber from oat grain and applying a food-grade depolymerization process to shorten the polysaccharide chain length of the fiber. BG-OS retains the fiber structure of oat fiber but has a shorter chain length, which makes it water soluble and easily formulated into any food.
  Other Names: Oat beta-glucan oligosaccharides
  Arms: 10 g/day of oat fiber; 20 g/day of oat fiber

SUMMARY:
The goal of this interventional study is to evaluate the tolerability and potential health benefits of oat fiber oligosaccharide (BG-OS) in healthy adults aged 18-70 years.

The main questions it aims to answer are:

* Does oat fiber dose impact gastrointestinal tolerability, as assessed by changes in symptoms using the Gastrointestinal Symptom Rating Scale (GSRS)?
* Does oat fiber reduce postprandial glucose levels after a white rice challenge? Researchers will compare three groups receiving different doses of oat fiber (5 g, 10 g, and 20 g) to assess dose-related effects.

Participants will:

* Complete daily surveys on gastrointestinal symptoms, diet, energy, and sleep quality.
* Use a continuous glucose monitoring device (CGM) to track glucose levels throughout the study.
* Participate in standardized white rice challenge tests to measure glucose uptake during baseline and at one time point during study.
* Provide stool samples during baseline and at the end of the study for gut microbiota analysis.
* Undergo blood tests for biomarkers like CBC, CMP, and A1C at the beginning and end of the study.

DETAILED DESCRIPTION:
The rationale for this study is to determine the gastrointestinal tolerability of a food-grade fiber obtained from oat (BG-OS) in healthy participants. Additionally, the study aims to observe the effects of the BG-OS on glucose uptake (as measured by Continuous Glucose Monitors or CGM) after a dietary challenge with cooked white rice, other potential health benefits of oat, and gut microbiota via activities and technologies that can successfully and effectively be completed and utilized in a home setting.

Outcomes will be examined in a broad age-range of adults who have chosen to try these products. The study incorporates participant reported outcomes and surveys, the use of a CGM device and carbohydrate (white rice) dietary challenge tests, at-home stool collection and standard blood sample collection for complete blood count (CBC), comprehensive metabolic panel (CMP) tests, and A1C hemoglobin test.

ELIGIBILITY:
Inclusion Criteria:

* Age: Healthy adults aged 18 to 70 years.
* Language Proficiency: Able to read and understand English.
* Informed Consent: Capable of providing informed consent.
* Technology Access: Must have a personal smartphone device.
* Able to download an app
* Study Commitment: Willing and able to complete all study assessments over a period of up to 7 weeks.

Exclusion Criteria:

* Technology Access: Lack of a smartphone and/or internet access.
* Medical Conditions:

Significant abnormal laboratory values (CBC, CMP, or A1C ≥ 6.5%) at screening.

Diagnosed with gastrointestinal, digestive, or metabolic diseases, including:

Crohn's disease Ulcerative colitis Irritable bowel syndrome Celiac disease Gluten allergy Diabetes Obesity Significant illness, disease, or condition that may interfere with study participation or outcomes, as determined by the principal investigator.

* Allergies: Known allergic reactions to any component of the study product or rice challenge product.
* Medications: Prescribed medications likely to influence study measures.
* Diet and Supplements:

Use of fiber supplements within 30 days prior to enrollment or during the study.

Major changes in diet or exercise 30 days prior to enrollment or during the study.

* Antibiotics Use: Use of antibiotics within 30 days prior to enrollment or during the study.
* Pregnancy and Breastfeeding: Pregnant, planning to become pregnant, or currently breastfeeding.
* Substance Use: Excessive alcohol use or substance abuse.
* Compliance Concerns: Unlikely to comply with the study protocol for any reason, as determined by the principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | On day 5, day 12 and day 19
  Change in gastrointestinal symptoms as measured by mean total score on the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS comprises 15 items, each rated on a Likert scale from 1 (no discomfort) to 7 (severe discomfort). Higher total scores indicate worse gastrointestinal symptoms

SECONDARY OUTCOMES:
Change in Postprandial Glucose Uptake after a white rice challenge (iAUC) | Day 3 (baseline), Day 6 (after first use of study product), Day 12 (after 1 week of use of study product), and Day 19 (end of intervention, after 2 weeks of use of study product).
  Change in postprandial glucose uptake measured by incremental Area Under the Curve (iAUC) using data from a Continuous Glucose Monitoring (CGM) device.
Change in Postprandial Glucose Uptake after a white rice challenge (Peak Glucose levels) | Day 3 (baseline), Day 6 (after first use of study product), Day 12 (after 1 week of use of study product), and Day 19 (end of intervention, after 2 weeks of use of study product).
  Change in peak glucose levels measured using a Continuous Glucose Monitoring (CGM) device.

OTHER OUTCOMES:
Glucose uptake dynamics | During baseline and throughout product use period (From Day 1 up to day 19)
  Changes in glucose uptake dynamics as measured by a CGM device
Effect on appetite, anxiety, mood | Day 5 (baseline), Day 12 (after 1 week of use of study product), and Day 19 (end of intervention, after 2 weeks of use of study product).
  Changes measured by weekly questionnaire that consists of 12 questions on appetite, anxiety and mood.
Gastrointestinal symptoms, sleep quality, energy levels, change in diet | Daily at baseline and daily throughout product use period (from Day 1 up to Day19)
  Changes measured by daily questionnaire that consists of 5 questions on participant experience of change in diet, energy levels and sleep quality.
Gut microbial composition | Once during baseline period (Day 1 to Day 5) and once at the end of study product use (Day 18 to Day 22)
  Changes in gut microbiota composition as analyzed by relative abundance of bacterial taxa in the stool samples
Gut microbial function | Once during baseline period (Day 1 to Day 5) and once at the end of study product use (Day 18 to Day 22)
  Changes in gut microbiota function as analyzed by quantification of key microbial-derived short chain fatty acids in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, M.D., Ph.D., Principal Investigator — People Science, Inc.
Locations (1):
- People Science Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No